CLINICAL TRIAL: NCT01097317
Title: NMES for Patients With NSCLC Receiving Palliative Chemotherapy. Is Neuromuscular Electrical Stimulation an Acceptable and Feasible Supportive Therapy for Patients With Non-Small Cell Lung Cancer Receiving Palliative Chemotherapy?
Brief Title: First-Line Chemotherapy With or Without Neuromuscular Electrical Stimulation in Treating Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000669234; WCTU-NMES; ISRCTN-42944026; EU-21019; NCRI-LCSUPAC-35
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2010-09

CONDITIONS: Chemotherapeutic Agent Toxicity; Fatigue; Lung Cancer; Musculoskeletal Complications
Keywords: chemotherapeutic agent toxicity; musculoskeletal complications; fatigue; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Fatigue; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Vinorelbine; Therapeutics

INTERVENTIONS:
Drug: carboplatin
Drug: vinorelbine tartrate
Other: neuromuscular electrical stimulation
Other: physiologic testing
Procedure: fatigue assessment and management
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemotherapy can lead to a loss of leg muscle strength. Neuromuscular electrical stimulation may improve muscle strength and quality of life. It is not yet known whether chemotherapy given together with neuromuscular electrical stimulation is more effective than chemotherapy alone in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying first-line chemotherapy given together with neuromuscular electrical stimulation to see how well it works compared with chemotherapy alone in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of first-line palliative chemotherapy alone versus palliative chemotherapy in combination with neuromuscular electrical stimulation (NMES) in patients with non-small cell lung cancer.

Secondary

* To determine if NMES is safe for patients undergoing palliative chemotherapy.
* To determine to what extent 3 or 4 courses of palliative chemotherapy impact leg muscle strength, body composition, and physical activity levels and if the use of NMES influence these changes.
* To determine the rate of recovery or decline in leg muscle strength, body composition, and physical activity levels following completion of 3 or 4 courses of palliative chemotherapy and if the use of NMES influences these changes.
* To assess patient attitudes to the use of NMES during palliative chemotherapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive first-line palliative chemotherapy comprising carboplatin and vinorelbine in weeks 1, 4, 7, and 10 as part of usual care at Nottingham University Hospital National Health Service Trust.
* Arm II (experimental): Patients receive chemotherapy as in arm I. Patients also undergo, at home, neuromuscular electrical stimulation (NMES) in weeks 2-12 (to the anterior thighs) 3 times a week for 30 minutes. NMES treatment increases in duration on a weekly basis from 11% to 18% to 25%, and then remaining constant thereafter.

All patients undergo assessment of quadriceps muscle strength, body composition, physical activity level, nutritional intake, and fatigue at baseline and week 9, and week 17 or 20. Patients complete quality-of-life questionnaires (EORTC-C30 and LC-13) at baseline, at week 9, and at week 17 or 20.

After completion of study treatment, patients are followed up for 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer
* Scheduled to receive 3 or 4 courses of first-line palliative chemotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Not pregnant or nursing
* Able to use neuromuscular electrical stimulation device
* No implanted cardiac pacemaker
* No epilepsy
* No spinal cord pathology

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to neuromuscular electrical stimulation (NMES) therapy

SECONDARY OUTCOMES:
Safety of NMES
Quadriceps muscle strength
Body composition
Physical activity level
Nutritional intake
Fatigue
Quality of life using the EORTC-C30 and LC-13 questionnaire
Overall objective clinical response to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilcock, MD, Principal Investigator — Nottingham City Hospital
Locations (1):
- Nottingham City Hospital, Nottingham, England, United Kingdom